CLINICAL TRIAL: NCT06086457
Title: PD-1 Inhibitor Plus Chemotherapy With or Without Radiotherapy in Patients With Metastatic Esophageal Cancer: A Randomized Multicenter Phase III Trial
Brief Title: PD-1 Inhibitor Plus Chemotherapy With or Without Radiotherapy in Patients With Metastatic Esophageal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Beijing Cancer Prevention & Treatment Society (Other); Hebei Medical University Fourth Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Fujian Cancer Hospital (Other Government); Anyang Tumor Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Sichuan Cancer Hospital and Research Institute (Other); Tengzhou Central People's Hospital (Other Government); The First Affiliated Hospital of Xiamen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); Changzhou Cancer Hospital of Soochow University (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEIR 0
Record Dates: First submitted 2023-09-21; First posted 2023-10-17 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Neoplasms
Keywords: Radiotherapy; PD-1 inhibitor
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiation; Drug Therapy; Immune Checkpoint Inhibitors; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 inhibitor plus chemotherapy arm (Active Comparator): Drugs: TP or PF regimen depended on investigator's choice. A maximum of six cycles was recommended for chemotherapy.
  Biological: PD-1 inhibitor (Camrelizumab).
  Interventions: Drug: TP or PF regimen depended on investigator's choice.; Biological: PD-1 inhibitor
- Radiotherapy arm (Experimental): Radiation: Intensity-modulated Radiation Therapy/Volumetric Modulated Arc Therapy (IMRT/VMAT) technique. Patients will receive radiotherapy between the first and third cycle of chemotherapy.
  Drugs: TP or PF regimen depended on investigator's choice. Biological: PD-1 inhibitor (Camrelizumab).
  Interventions: Radiation: Radiation; Drug: TP or PF regimen depended on investigator's choice.; Biological: PD-1 inhibitor

INTERVENTIONS:
Radiation: Radiation — IMRT/VMAT technique. Patients receive radiotherapy once daily, 5 days a week for an average of 5 weeks. Radiotherapy is delivered to achieve a dosage of 50Gy in 25 fractions to planning gross tumor volume (PGTV) with involved site included.
  Other Names: Modern intensity modulated radiotherapy
  Arms: Radiotherapy arm
Drug: TP or PF regimen depended on investigator's choice. — A maximum of six cycles was recommended for chemotherapy. Chemotherapy Regimen 1(TP regimen A): Nab-paclitaxel(Albumin-bound paclitaxel) 110-130mg/ m2，d1，d8; Cisplatin 60-75mg/ m2，d1；Q3W； Chemotherapy Regimen 2 (TP regimen B): Paclitaxel 150-175 mg/m2, d1; Cisplatin 60-75mg/ m2，d1；Q3W； PD-1 inhibitor 200mg, d1, Q3W Chemotherapy Regimen 3 (PF regimen): Capecitabine 800mg/m2, bid, d1-14; Cisplatin 25-30mg/m2, d1,d2, Q3W.
  Other Names: Chemotherapy
Biological: PD-1 inhibitor — Camrelizumab (200mg, d1, Q3W) was continued until disease progression, unacceptable toxicity, death, physician or patient decision to withdraw, non-compliance, or discontinuation for administrative reasons (up to 35 cycles).
  Other Names: Camrelizumab

SUMMARY:
The treatment efficacy for stage IVb esophageal cancer has been improved through chemotherapy combined with immunotherapy recently.

On this basis, the investigators intend to conduct a prospective, multicenter phase III clinical trial to assess whether radiotherapy with concurrent chemotherapy and immunotherapy could further improve the survival of patients with metastatic esophageal cancer.

Accompanied tissue samples, blood samples and urine samples will be analyzed by molecular biological detection (Including Whole Exome Sequencing and proteomics) to explore potential biomarkers for predicting outcomes, efficacy and toxicity.

DETAILED DESCRIPTION:
Esophageal cancer (EC) is one of the most common carcinomas with high morbidity and mortality worldwide. More than 30% of the patients were stage IV when diagnosed. Fluoropyrimidine plus platinum-based chemotherapy is recommended as first-line treatment for patients with metastatic EC for approximately four decades, however, only minimal improvement has been reached in overall survival (OS).

Recently, immune checkpoint inhibitors have shown effective antitumor activity in patients with unresectable, advanced or metastatic EC. Several randomized trials have demonstrated the PD-1 inhibitor could further improve the OS in patients with advanced esophageal squamous cell carcinoma (ESCC) on the basis of chemotherapy. Chemotherapy combined with immunotherapy has become one of the the standard treatment modality for advanced EC.

As reported, for the patients with metastatic lung cancer or EC, locoregional radiotherapy could improve survival. However, high-level evidence is still needed to assess whether these patients can benefit from local radiotherapy.

The efficacy of immunotherapy combined with chemotherapy is obviously better than that of chemotherapy alone. On this basis, locoregional radiotherapy may help some patients with advanced EC improve local control, relieve the local symptoms and improving the quality of life.

Therefore, the investigators intend to conduct a prospective, multicenter phase III trial to assess the efficiency and safety of radiotherapy with chemotherapy and immunotherapy of patients with metastatic EC. Accompanied tissue samples, blood samples and urine samples will be analyzed by molecular biological detection to explore potential biomarkers for predicting outcomes, efficacy and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥18 years, any gender
* 2. Histologically or cytologically confirmed squamous cell carcinoma of esophageal cancer. The initial clinical stage is IVb (2018 American Joint Committee on Cancer (AJCC) Cancer Staging Manual, 8th Edition) , with distant metastasis involving no more than 2 organs (lymph node metastasis is counted);
* 3. ECOG (Eastern Cooperative Oncology Groupper) formance status <= 1. Patients aged 65 years and over need to complete G8 screening or Comprehensive Geriatric Assessment, and the final evaluation is good;
* 4.There was no significant abnormality in laboratory routine indicators such as blood routine and liver and kidney function;
* 5.No prior history of thoracic radiation;
* 6.Expected survival is more than 12 weeks;
* 7.Informed consent provided.

Exclusion Criteria:

* 1.Patients with other cancer history except hypopharyngeal carcinoma in situ, non-malignant skin cancer and cervical carcinoma in situ.
* 2.Received surgery (except ostomy), chemotherapy or other anti-tumor treatment before enrollment；
* 3. Active infection currently exists . The following conditions occurred within 6 months before randomization: myocardial infarction, cerebrovascular accident, or received gastrointestinal, neurological, cardiopulmonary surgery;
* 4. History of allergy to chemotherapy drugs or autoimmune disease;
* 5. Participate in other clinical trials at present or within 4 weeks before enrollment;
* 6.There are factors such as high risk of fistula that radiotherapy cannot be safely carried out as assessed by the radiation oncologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identity
Enrollment: 436 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2029-08-28 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 33 months (through Primary Analysis cut-off date of 30-May-2026).
  Overall survival was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS is reported for all participants of the Intent-To-Treat (ITT) population (all randomized).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 33 months (through Primary Analysis cut-off date of 30-May-2026).
  PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 as assessed by the investigator, or death due to any cause, whichever occurred first.
Objective Response Rate (ORR) | Up to approximately 33 months (through Primary Analysis cut-off date of 30-May-2026).
  ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. as assessed by the investigator.
Acute toxicity Rate | One month within the end of one specific treatment.
  Acute toxicity rate was defined as the frequency of toxicities related to the treatment, which arises within one month after administration, according to National Cancer Institute Common Terminology Criteria for Adverse Event,Version 5.0 (CTC Adverse Event 5.0).
Late toxicity rate | One month after the end of one specific treatment.
  Late toxicity rate was defined as the frequency of toxicities related to the treatment, which arises after one month after administration, according to National Cancer Institute Common Terminology Criteria for Adverse Event,Version 5.0 (CTC Adverse Event 5.0).
QUALITY OF LIFE: Change From Baseline in the EORTC QLQ-C30 Subscale Score in Participants | 24 months
  The score of the participants evaluated by The EORTC core quality of life questionnaire (QLQ-C30) . The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score represents a higher response level. Thus a high score for a functional scale represents a high/healthy level of functioning.
QUALITY OF LIFE: Change From Baseline in the EORTC QLQ-OES18 Subscale Score in Participants | 24 months
  The score of the participants evaluated by The EORTC Quality of Life Questionnaire - Oesophageal Cancer Module (EORTC QLQ-OES18). The EORTC QLQ-OES18 is a disease-specific questionnaire developed and validated to address measurements specific to esophageal cancer and contains 18 items assessing symptoms of dysphagia, pain, reflux symptoms, eating restrictions, anxiety, dry mouth, taste, body image, and hair loss. All subscale items were scored using a four-point Likert scale with the following response choices: 1=not at all, 2=a little, 3=quite a bit, 4=very much. Raw scores for the subscales were standardized into a range of 0 to 100 by linear transformation, with higher symptom scores represent a higher ("worse") level of symptoms.

OTHER OUTCOMES:
Biomarkers for the predicting of efficacy | 33 months
  To explore the dynamic changes of circulating tumor DNA (the frequency of specific mutations by Next-generation sequencing Methodology) from baseline, before and after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Wen-Yang Liu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital, CAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in esophageal cancer. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact liuwenyang@cicams.ac.cn

REFERENCES:
- [Background] Sun JM, Shen L, Shah MA, Enzinger P, Adenis A, Doi T, Kojima T, Metges JP, Li Z, Kim SB, Cho BC, Mansoor W, Li SH, Sunpaweravong P, Maqueda MA, Goekkurt E, Hara H, Antunes L, Fountzilas C, Tsuji A, Oliden VC, Liu Q, Shah S, Bhagia P, Kato K; KEYNOTE-590 Investigators. Pembrolizumab plus chemotherapy versus chemotherapy alone for first-line treatment of advanced oesophageal cancer (KEYNOTE-590): a randomised, placebo-controlled, phase 3 study. Lancet. 2021 Aug 28;398(10302):759-771. doi: 10.1016/S0140-6736(21)01234-4. PMID 34454674
- [Background] Luo H, Lu J, Bai Y, Mao T, Wang J, Fan Q, Zhang Y, Zhao K, Chen Z, Gao S, Li J, Fu Z, Gu K, Liu Z, Wu L, Zhang X, Feng J, Niu Z, Ba Y, Zhang H, Liu Y, Zhang L, Min X, Huang J, Cheng Y, Wang D, Shen Y, Yang Q, Zou J, Xu RH; ESCORT-1st Investigators. Effect of Camrelizumab vs Placebo Added to Chemotherapy on Survival and Progression-Free Survival in Patients With Advanced or Metastatic Esophageal Squamous Cell Carcinoma: The ESCORT-1st Randomized Clinical Trial. JAMA. 2021 Sep 14;326(10):916-925. doi: 10.1001/jama.2021.12836. PMID 34519801
- [Background] Guttmann DM, Mitra N, Bekelman J, Metz JM, Plastaras J, Feng W, Swisher-McClure S. Improved Overall Survival with Aggressive Primary Tumor Radiotherapy for Patients with Metastatic Esophageal Cancer. J Thorac Oncol. 2017 Jul;12(7):1131-1142. doi: 10.1016/j.jtho.2017.03.026. Epub 2017 Apr 28. PMID 28461255